CLINICAL TRIAL: NCT01547559
Title: Evaluation of Preventive and Treatment Effects of Hp Eradication and Teprenone in Patients Taking NSAIDs
Brief Title: Research for Prevention and Treatment of NSAIDs Related Gastrointestinal Side Effects
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Xinxin Huang, doctor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 5010-2007005
Record Dates: First submitted 2012-03-07; First posted 2012-03-08 (Estimated); Last update posted 2014-10-21 (Estimated); Status verified 2014-10

CONDITIONS: Non-steroidal Anti-inflammatory Drug Adverse Reaction

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (7):
- part1:blank control (No Intervention): NO maintain drugs with Hp negative patients.
- part1:teprenone 1 (Experimental): maintain treatment with Teprenone for Hp negative patients
  Interventions: Drug: part1:teprenone
- part1:EAC-T (Experimental): eradication of Hp with triple treatment
  Interventions: Drug: part1:EAC-T
- part1：EA-EMC-T (Experimental): eradication of Hp with sequential therapy
  Interventions: Drug: part1:EA-EMC-T
- part1：T-T (Active Comparator): Teprenone as maintain drugs for Hp positive patients
  Interventions: Drug: part1:teprenone
- part2:GGA group (Experimental): Geranylgeranylacetone plus diclofenac sodium for patients with rheumatic diseases
  Interventions: Drug: part2:GGA group
- part2:control group (No Intervention): diclofenac sodium only for patients with rheumatic diseases

INTERVENTIONS:
Drug: part1:teprenone — Teprenone 50mg tid after meal for Hp negative patients.
  Other Names: teprenone treatment
  Arms: part1:teprenone 1
Drug: part1:EAC-T — esomeprazole 20 mg, amoxicillin 1 g, and clarithromycin 500 mg, each twice daily followed by gastric mucosal protective therapy with teprenone 50mg three times daily for 11 weeks
  Other Names: EAC-T treatment
  Arms: part1:EAC-T
Drug: part1:EA-EMC-T — esomeprazole 20 mg plus amoxicillin 1 g, twice daily for 5 days, then esomeprazole 20 mg with clarithromycin 500 mg and metronidazole 500 mg, twice daily for another 5 consecutive days) followed by teprenone 50mg three times daily until 12 weeks
  Other Names: EA-EMC-T treatment
  Arms: part1：EA-EMC-T
Drug: part1:teprenone — Teprenone 50mg tid after meal for Hp positive patients.
  Other Names: T-T treatment
  Arms: part1：T-T
Drug: part2:GGA group — GGA 50mg three times daily plus diclofenac sodium 75mg once a day for patients with rheumatic diseases.
  Other Names: GGA
  Arms: part2:GGA group

SUMMARY:
We aim to evaluate the protective effects of eradication of HP and continue using Geranylgeranylacetone (GGA) on NSAIDs related gastroenterological lesions. We further aim to explore the effect of GGA on small-intestinal mucosal injuries induced by diclofenac sodium in patients with rheumatic diseases who didn't take NSAIDs in the preceding 6 months.

DETAILED DESCRIPTION:
NSAIDs are mainly used drugs in rheumatic disease and cardiologic disease. However the gastroenterological lesions prevent patients get benefits from continuing taking NSAIDs. HP is another important factor that increase gastroenterological lesions. Both HP and NSAIDs increase risk of peptic ulcers, however, no exact relation between these two factors has been found. It is important to evaluate the protective effects of eradication of HP in NSAIDs-taking patients. In many countries ,PPI is recommended as maintain treatment in NSAIDs-taking patients to prevent gastroenterological lesions. A multicenter, open-label, randomized, parallel-group study is needed to prove the effects of Teprenone as a replacer of PPI in maintain treatment.On the other hand, Small-intestinal mucosal injuries induced by non-steroidal anti-inflammatory drugs (NSAIDs) are common. However, there are still no effective and reliable interventions established. Geranylgeranylacetone (GGA) is a mucosal protective agent, so we develop an additional trail to clarify the discrepancies of GGA effects on NSAIDs-induced small-intestinal mucosal injuries.

ELIGIBILITY:
part1:

Inclusion Criteria:

1. informed consents be given before treatment
2. NSAIDs taking patients
3. not taking PPI or other digestive drugs during previous 1 months
4. age ranging from 18～80 years old

Exclusion Criteria:

1. having any severe acute or chronic complications
2. renal dysfunction, blood creatinine≥150µmol/L
3. blood aminotransferase level rising up(more than 2 times of the normal level)
4. any severe cardiac disease including congestive cardiac failure, unstable angina and myocardial infarct in 12 months
5. serious hypertension (systolic pressure≥180mmHg and/ or diastolic pressure≥110mmHg)
6. chronic or acute pancreatic disease
7. severe systematic diseases or malignant tumor
8. allergic to the drugs using in the trial
9. any factors interfering the result
10. female patients incline to be pregnant
11. being treated with drugs influencing gastroenterological conditions.
12. poor compliance part2:

Inclusion Criteria:

1.18 to 65 years of age 2.patients with rheumatic diseases such as ankylosing spondylitis , rheumatoid arthritis and undifferentiated arthritis 3.planning to take diclofenac sodium for at least 12 weeks 4.having freely been given their fully informed consent based on their full understanding

Exclusion Criteria:

1. Patients were excluded if they had a history of peptic ulcer or gastrointestinal bleeding
2. had serious liver, kidney, heart, or lung disease
3. had suspected small-bowel obstruction
4. had a history of gastrointestinal surgery except for appendectomy
5. had a drug addiction or alcoholism; were pregnant or hoped to become pregnant during the study period
6. were taking anti-secretory drugs such as PPIs or H2 receptor antagonists (H2RA), or other gastric mucosal protective drugs
7. had a lack of consent to the surgery required if the capsule endoscope was retained in the body
8. were judged to be inappropriate for this study by the investigator

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 369 (Actual)
Dates: Start 2007-06; Primary Completion 2014-11 (Estimated)

PRIMARY OUTCOMES:
part1:the total proportion of peptic ulcers after treatment | 12 weeks
part2:Capsule endoscopy findings of small-intestinal mucosal injuries after treatment | 12 weeks

SECONDARY OUTCOMES:
part1:the development of gastroduodenal ulcers | 12 weeks
part1:the healing rate of gastroduodenal ulcers | 12 weeks
part1:the improvement of erosions | 12 weeks
part2：capsule endoscopy (CE) Lewis Score after treatment | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Minhu Chen, MD PHD, Study Chair — First Affiliated Hospital, Sun Yat-Sen University
Locations (1):
- the first Affiliated Hospital of Sun Yat-Sen university, Guangzhou, Guangdong, China

REFERENCES:
- [Derived] Xiong L, Huang X, Li L, Yang X, Liang L, Zhan Z, Ye Y, Chen M. Geranylgeranylacetone protects against small-intestinal injuries induced by diclofenac in patients with rheumatic diseases: a prospective randomized study. Dig Liver Dis. 2015 Apr;47(4):280-4. doi: 10.1016/j.dld.2015.01.005. Epub 2015 Jan 20. PMID 25660821